CLINICAL TRIAL: NCT02438072
Title: Cocktail Phenotypic Approach to Explore Antidepressant Pharmacokinetic Variability: a Pilot Study
Brief Title: Drug Metabolism and Antidepressant
Acronym: METADEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Celia Lloret-Linares, Doctor, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CER-14051
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Depression
Keywords: antidepressive agent; drug metabolism; CYP450; P-glycoprotein; Phenotypic study
MeSH Terms: conditions — Depression | interventions — Omeprazole; Flurbiprofen; Dextromethorphan; Midazolam; fexofenadine; Bupropion; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall population (Other)
  Interventions: Drug: Omeprazole (10 mg, A02BC01)

INTERVENTIONS:
Drug: Omeprazole (10 mg, A02BC01) — The cocktail of drug substrates will be given one time, one day during the study, to explore the activity of CYP 1A2, 2B6, 2C9, 2C19, 3A4, 2D6, and the P-gp
  Other Names: Flurbiprofen (10 mg, M01AE09); Dextromethorphan (10 mg, R05DA09); Midazolam (1 mg, N05CD08); Fexofenadine (25mg, R06AX26 ); Bupropion (20 mg, N06AX12); Caffeine (50 mg, N06BC01)

SUMMARY:
We propose here to explore systematically the association between drug-metabolizing enzymes activity assessed by a phenotypical approach and antidepressant plasma concentration, efficacy and tolerance in the clinical setting. During one year, patients receiving antidepressant will be included in tis prospective clinical, naturalistic and descriptive pilot study.

DETAILED DESCRIPTION:
* Objectives To describe drug metabolism variability in depressive patients using a phenotypic approach
* Study design Prospective, clinical, naturalistic, descriptive study During a consultation with their clinician, depressive patients will receive information.

During the visit V0 with an investigator: patients will be included:

* Verification of inclusion and non inclusion criteria
* Reminder participation conditions
* Inclusion, signature of consent
* Collection of clinical and demographic features Between V0 and V1, for patients with change in antidepressant therapy, will take place telephone interviews every two weeks, conducted by the clinician to evaluate treatment depression response (tolerance and efficacy)

During the visit V1, will take place:

* Phenotypic study
* Genetic study
* Dosage of current antidepressant drug
* Clinical evaluation: efficacy and tolerance

  * Number of patients During one year, the protocol will be proposed to all patients with depression and decision of change in antidepressant therapy, and all patients with stability od prescription since almost 6 weeks. The inclusion of approximately 100 patients is expected.
  * Name of the finished product Zyban®, Froben®, Antra®, Bexine®, Dormicum® Telfast®
  * Name of the active substance Omeprazole (10 mg, A02BC01) Caffeine (50 mg, N06BC01) Flurbiprofen (10 mg, M01AE09) Dextromethorphan (10 mg, R05DA09) Midazolam (1 mg, N05CD08) Fexofenadine (25mg, R06AX26 ) Bupropion (20 mg, N06AX12)
  * Duration of treatment One time during the study, one day (Visit 1)
  * Time plan of research -Duration for the patient: The study will stop when the patient has performed the V1 study Minimal delay between V0 and V1: 6 weeks (5-7 weeks) : for patient with decision to change the treatment, 5 days for patients with stability of treatment since almost 6 weeks.

Maximal delay of participation for the patient: 4 months even when V1 was not performed

-Overall duration of inclusion: one year Maximal overall duration of the study: 12 months+4 months= 16 months Maximal duration for the analytical study since the beginning of the study= 16 months+6 months: 22 months.

Maximal delay for communication of the results: 2 years after the beginning of the study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical diagnosis of depression and decision to change antidepressant therapy (augmentation or switch) OR Patients with clinical diagnosis of depression and stability of prescription since almost 6 weeks
2. Male and female aged from 18 to 70 years
3. Volunteers to participate to the study
4. Understanding of French language and able to give a written inform consent.

Exclusion Criteria:

Renal or hepatic impairment (Clearance below 60mL/min, AST or ALT over 3N) Sensitivity to any of the substrate drugs used ECG showing long QT interval (>0.46sec) No antidepressant dosage available Current pregnancy or desire to get pregnant

Criteria to perform V1 Sufficient compliance between V0 and V1 Six weeks period without change in antidepressant therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
CYP1A2 activity | >two hours after an oral intake of the cocktail probe drugs
  paraxanthine/caffeine
CYP2B6 activity | >two hours after an oral intake of the cocktail probe drugs
  4-hydroxybupropion/ bupropion
CYP2D6 activity | >two hours after an oral intake of the cocktail probe drugs
  dextrorphan / dextromethorphan
CYP2C9 activity | >two hours after an oral intake of the cocktail probe drugs
  4-hydroxyflurbiprofen/ flurbiprofen
CYP2C19 activity | >two, three and six hours after an oral intake of the cocktail probe drugs
  5-hydroxyomeprazole/ omeprazole
CYP3A4 activity | >two hours after an oral intake of the cocktail probe drugs
  1-hydroxymidazolam/ midazolam
P-gp activity | >two, three and six hours after an oral intake of the cocktail probe drugs
  Limited sampling fexofenadine AUC

SECONDARY OUTCOMES:
Antidepressant Concentration | almost 6 weeks after the last treatment change
Antidepressant tolerance | almost 6 weeks after the last treatment change
  FISBER test
Antidepressant efficacy | almost 6 weeks after the last treatment change
  Tests: MADRS, Hamilton, QIDS-16

CONTACTS AND LOCATIONS:
Overall Officials: Celia Lloret-Linares, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Background] Bosilkovska M, Samer CF, Deglon J, Rebsamen M, Staub C, Dayer P, Walder B, Desmeules JA, Daali Y. Geneva cocktail for cytochrome p450 and P-glycoprotein activity assessment using dried blood spots. Clin Pharmacol Ther. 2014 Sep;96(3):349-59. doi: 10.1038/clpt.2014.83. Epub 2014 Apr 10. PMID 24722393
- [Result] Hall-Flavin DK, Winner JG, Allen JD, Carhart JM, Proctor B, Snyder KA, Drews MS, Eisterhold LL, Geske J, Mrazek DA. Utility of integrated pharmacogenomic testing to support the treatment of major depressive disorder in a psychiatric outpatient setting. Pharmacogenet Genomics. 2013 Oct;23(10):535-48. doi: 10.1097/FPC.0b013e3283649b9a. PMID 24018772
- [Derived] Lloret-Linares C, Bosilkovska M, Daali Y, Gex-Fabry M, Heron K, Bancila V, Michalopoulos G, Perroud N, Richard-Lepouriel H, Aubry JM, Desmeules J, Besson M. Phenotypic Assessment of Drug Metabolic Pathways and P-Glycoprotein in Patients Treated With Antidepressants in an Ambulatory Setting. J Clin Psychiatry. 2018 Mar/Apr;79(2):16m11387. doi: 10.4088/JCP.16m11387. PMID 29570971